CLINICAL TRIAL: NCT05754502
Title: Observational Study of Effectiveness and Safety of Trastuzumab Emtansine (T-DM1) in HER2-positive Breast Cancer Patients With Residual Invasive Disease Following Neoadjuvant Chemotherapy and Anti-HER2 Target Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Consorzio Oncotech (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: GIM26-TRASTHER
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Trastuzumab emtansine — observational study. After the signature of the Informed Consent Form, all their data reported in the medical charts up to then (as detailed in section 12 of the protocol) will be extracted retrospectively and inserted in the study database. From the end of the washout period following the last treatment with T-DM1, each subject will enter in an observation phase for a maximum of 3 years, or until death whichever happens first. This phase will be prospective after the signature of the Informed Consent Form.

SUMMARY:
This is an observational, multi-centre study analysing data from patients treated with T-DM1 within the compassionate use program AL41711. During the compassionate use program AL41711, subjects received T-DM1 treatment for a total of 14 cycles or less, in case of disease recurrence or unmanageable toxicity. After the completion of the treatment, and 90 days of wash-out period, they can be enrolled in the study. After the signature of the Informed Consent Form, all their data reported in the medical charts up to then (as detailed in section 12 of the protocol) will be extracted retrospectively and inserted in the study database. From the end of the washout period following the last treatment with T-DM1, each subject will enter in an observation phase for a maximum of 3 years, or until death whichever happens first. This phase will be prospective after the signature of the Informed Consent Form.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Patients who have received T-DM1 treatment within the compassionate use program AL41711 and have completed the entire treatment for at least 90 days or have interrupted it prematurely, due to disease recurrence or unmanageable toxicity, for at least 90 days, corresponding to the wash out period;

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include approximately 300 patients with HER2-positive breast cancer that do not reach a pathological complete response following neoadjuvant chemotherapy and anti-HER2 target therapy and received T-DM1 within the compassionate use program AL41711.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2024-09-21 (Estimated); Study Completion 2025-05-02 (Estimated)

PRIMARY OUTCOMES:
Complete response-Effectiveness of treatment with T-DM1 | up to 36 months
  assess the long term effectiveness of treatment with T-DM1 as compassionate use in patients with HER2-positive breast cancer that do not reach a complete response following neoadjuvant chemotherapy and anti-HER2 target therapy

CONTACTS AND LOCATIONS:
Locations (28):
- Italy (28):
  - Nuovo ospedale di Prato - S. Stefano, Prato, Firenze
  - A.O.U. Ospedali Riuniti Umberto I, Ancona
  - IRCCS Istituto Tumori "Giovanni Paolo II", Bari
  - Humanitas Centro Catanese di Oncologia U.O. Oncologia Medica, Catania
  - Azienda Ospedaliera Istituti Ospitalieri di Cremona, Cremona
  - I.R.C.C.S. A.O.U San Martino - IST, Genova
  - ASST Lecco - P.O. "A. Manzoni", Lecco
  - Istituto Europeo di Oncologia, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - A.O.U Policlinico di Modena, Modena
  - Azienda Ospedaliera dei Colli - P.Monaldi, Napoli
  - Istituto Nazionale dei Tumori - Fondazione G. Pascale U.O. Oncologia Medica Senologica, Napoli
  - Università di Napoli Federico II - Facoltà di Medicina Dipartimento di Medicina Clinica e Chirurgia - Oncologia, Napoli
  - A.O.R.N. "A. Cardarelli", Napoli
  - A.O.U. 'Maggiore della Carità', Novara
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliera Universitaria di Parma - Oncologia Medica, Parma
  - Fondazione S. Maugeri IRCCS U.O. Oncologia Medica II, Pavia
  - A. O. U. Pisana - Ospedale S. Chiara, Pisa
  - IRCCS Arcispedale S.Maria Nuova, Reggio Emilia
  - Ospedale Sandro Pertini - ASL Roma 2, Roma
  - Fondazione Policlinico A. Gemelli, Roma
  - Fondazione Policlinico Gemelli, Roma
  - Policlinico Universitario Campus Biomedico, Roma
  - Istituto Clinico Humanitas Irccs, Rozzano
  - Azienda Ospedaliera 'San Giovanni di Dio e Ruggi D'Aragona' Struttura Complessa di Oncologia, Salerno
  - Ospedale Santa Chiara, Trento
  - ASST Sette Laghi - Ospedale Di Circolo e Fondazione Macchi, Varese

IPD SHARING:
Plan to Share IPD: No